CLINICAL TRIAL: NCT04975217
Title: Pilot Study Using Fecal Microbial Transplants in Patients With Pancreatic Cancer
Brief Title: Fecal Microbial Transplants for the Treatment of Pancreatic Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0788; NCI-2021-03484 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0788 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-05-25; First posted 2021-07-23 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Fecal Microbiota Transplantation; Parturition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (FMT, FMT capsules) (Experimental): Patients undergo FMT during colonoscopy. Patients also receive FMT capsules PO QW for 4 weeks in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care resection of tumor(s).
  Interventions: Procedure: Fecal Microbiota Transplantation; Drug: Fecal Microbiota Transplantation Capsule; Other: Questionnaire Administration; Procedure: Resection; Procedure: Therapeutic Colonoscopy

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — Undergo FMT
  Other Names: Fecal Material Transplantation; Fecal Transplantation; FMT; Poo Transplant; Poop Transplant; Stool Transplant
Drug: Fecal Microbiota Transplantation Capsule — Given PO
  Other Names: Fecal Microbiota Preparation Delivery Capsule; FMPCapDE; FMT Capsule DE; FMT Capsule Delivery; FMT DE Capsule
Other: Questionnaire Administration — Ancillary studies
Procedure: Resection — Undergo standard of care resection
  Other Names: Surgical Resection
Procedure: Therapeutic Colonoscopy — Undergo colonoscopy

SUMMARY:
This early phase I trial examines the safety and effects of fecal microbial transplants in treating patients with pancreatic cancer. scheduled for surgery to remove tumors. Fecal microbial transplant contains the normal microbes found in fecal (stool) material. Giving fecal microbial transplant may help control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety, tolerability, and feasibility of fecal microbiota transplantation (FMT) in resectable patients with pancreatic ductal adenocarcinoma (PDAC).

SECONDARY OBJECTIVES:

I. To assess changes in gut microbiome of PDAC patients after FMT. II. To assess changes in oral microbiome of PDAC patients after FMT. III. To assess changes in tumor microbiome of PDAC patients after FMT. IV. To determine immunological/molecular changes in the tumor after FMT.

OUTLINE:

Patients undergo FMT during colonoscopy. Patients also receive FMT capsules orally (PO) once weekly (QW) for 4 weeks in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care resection of tumor(s).

After completion of study treatment, patients are followed up at 2 weeks and 30, 60, 90, and 180 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are seen at MD Anderson Cancer Center
* Patients with pancreatic ductal adenocarcinoma (PDAC) diagnosis who are expected to have surgery (Whipple)
* Adequate hematological function, defined by white blood cell (WBC) count ≥ 3,000/microL, platelet count ≥75,000/microL, and Hgb ≥ 8 g/dL
* Adequate hepatic function defined by a total bilirubin level ≤ 1.5 × the upper limit of normal (ULN), an AST, level ≤ 2.5 × ULN, and an ALT level ≤ 2.5 × ULN
* Adequate renal function defined by an estimated creatinine clearance >30 mL/min according to the Cockcroft-Gault formula or by a creatinine clearance measurement from a 24-hour urine collection
* Age 18 years and above
* Male or female
* Willingness and ability to sign an informed consent
* Consent and ability to give blood and stool samples
* Consent to undergo a baseline core biopsy and colonoscopy for FMT delivery
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2

Exclusion Criteria:

* Age younger than 18 years
* Positive GI infection
* Patients with pancreatic cancer Stage T1N0
* Individuals at higher risk of colonization with MDROs
* Patient received antibiotics in the last 48 hours. Patients will be eligible to enroll if antibiotic therapy is discontinued for at minimum 48 hours prior to start of study
* Patients with active viral, bacterial or fungal infection
* History of inflammatory bowel disease, and/or radiation enteritis or colitis
* Pregnant and breastfeeding women
* Women of child-bearing potential who have positive urine or serum pregnancy test or refuse to do pregnancy test
* Has a diagnosis of immunodeficiency
* Peripheral WBC >12 x 10^9/L and/or temperature >38 degrees Celsius
* Subjects with neutropenia (ANC <1500)
* Swallowing dysfunction or known chronic aspiration
* Delayed gastric emptying
* History of intestinal obstruction
* Acute exacerbation of underlying comorbid condition
* Severely immunocompromised patients
* Allergies to drugs included as part of trial (antibiotics, loperamide or laxatives)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after surgery
  Will be measured by Common Terminology Criteria for Adverse Events, version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Florencia McAllister, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org